CLINICAL TRIAL: NCT04695327
Title: A Phase 1, Open-Label, Dose-escalation Clinical Trial of Tumor Necrosis Factor Alpha and Interleukin-2 Coding Oncolytic Adenovirus (TILT-123) in Patients With Injectable Solid Tumors
Brief Title: TNFα and IL-2 Coding Oncolytic Adenovirus TILT-123 Monotherapy
Acronym: TUNIMO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TILT Biotherapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILT-T115; 2020-001778-31 (EudraCT Number)
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor
Keywords: Oncolytic virus; Virotherapy; Immunotherapy; Adenovirus; TILT-123
MeSH Terms: conditions — Adenoviridae Infections | interventions — Tumor Necrosis Factor-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy (Experimental): Patients will receive multiple administrations of TILT-123.
  Escalation to the next dose of TILT-123 level will occur when the safety data has been evaluated for all patients in the preceding dose level.
  Interventions: Biological: TILT-123

INTERVENTIONS:
Biological: TILT-123 — TNFalpha and IL-2 coding oncolytic adenovirus TILT-123
  Other Names: TNFalpha and IL-2 coding oncolytic adenovirus TILT-123; Ad5/3-E2F-d24-hTNFa-IRES-hIL2

SUMMARY:
This is an open-label, phase 1, dose-escalation, multicenter trial evaluating the safety of oncolytic adenovirus TILT-123 as monotherapy in advanced solid tumor patients.

DETAILED DESCRIPTION:
This is an open-label, phase 1, dose-escalation trial evaluating the safety of TILT-123 as monotherapy in advanced solid tumor patients. TILT-123 is an oncolytic adenovirus coding for tumor necrosis factor alpha and interleukin 2. The trial includes 2 healthcare centers in Helsinki (Finland). Patients with different indications are expected to be treated in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent before any trial-related activities.
* Male or female over 18 years of age
* Pathologically confirmed refractory or recurrent injectable solid tumor, which cannot be treated with curative intent with available therapies.
* Standard therapy has failed, it does not exist, is not available or is unlikely to result in meaningful clinical benefit (as assessed by the investigator). Other appropriate evidence-based therapies have failed or are contraindicated.
* Multiple prior therapies (e.g. surgery, chemotherapy, checkpoint inhibitors, kinase inhibitors, biological therapies, hormonal therapies, radiation, etc) are allowed.
* At least one tumor (>14 mm in diameter) must be available for injections and biopsies for correlative analyses. The disease burden must be measurable, but does not need to fulfil RECIST 1.1.
* Adequate hepatic and renal functions as following:

  1. Platelets > 75 000/mm3
  2. Haemoglobin ≥ 100 g/L.
  3. AST and ALT < 3 x ULN.
  4. GFR >60 ml/min (Cockcroft-Gault formula).
  5. Leukocytes (WBC) > 3,0
  6. Bilirubin <1,5 x ULN 8. Men and women must be willing to use adequate forms of contraception from screening, during the trial, and for a minimum of 90 days after end of treatment, in accordance with the following:

  <!-- -->

  1. Women of childbearing potential: Barrier contraceptive method (i.e. condom) must be used in addition to one of the following methods: Intrauterine device or hormonal contraception (oral contraceptive pills, implant, transdermal patches, vaginal ring or long-acting injections).
  2. Women not of childbearing potential: Barrier contraceptive method (i.e. condom) must be used.
  3. Men: Barrier contraceptive method (i.e. condom) must be used.
* Demonstrated WHO/ECOG performance score of 0-1 at screening.
* Life expectancy time longer than 3 months.
* Capable of understanding and complying with parameters as outlined in the protocol.

Exclusion Criteria:

* Use of immunosuppressive medications (corticosteroids or drugs used in treatment of autoimmune disease). Exempted are the following which can be allowed at screening and during the trial: a) replacement corticosteroids if e.g. the patient has adrenal insufficiency after prior immunotherapy b) inhaled and topical treatments c) up to 20 mg per day of prednisone/prednisolone.
* Treated with any anti-cancer therapy within 30 days prior to the first virus injection. Anti-cancer therapy is defined as anti-cancer agents (e.g. cytotoxic chemotherapy, immunotherapy, signal-transduction inhibitors, etc) and investigational agents. An investigational agent is any drug or therapy that is currently not approved for use in humans. Continuation of hormonal therapy or use of bone modifying agents (eg. bisphosphonate or denosumab) is allowed if started at least 3 months before. Palliative radiation is not allowed within 14 days of the first virus injection (before or after), but it is allowed after day 15 during the trial treatment period, if deemed necessary by the investigator.
* Uncontrolled cardiac or vascular diseases.
* History of myocardial infarction or cerebral stroke within the previous 12 months before screening or is not sufficiently recovered from an older infarction or cerebral stroke.
* History of severe hepatic dysfunction, hepatitis or HIV.
* History of coagulation disorder.
* Any other medical condition or laboratory abnormality that in the judgment of the principal investigator, may increase the risk associated with study participation or may interfere with interpretation of study results and /or otherwise make the patient inappropriate for entry into this trial.
* Female patients who are pregnant, breastfeeding or intend to become pregnant.
* Untreated brain metastases. Treated brain metastases which have not progressed in 3 months prior to screening are allowed.
* Previously treated (within 5 years) with any oncolytic or replication deficient adenovirus.
* Allergy to ingredients present in the investigational medicinal products (ingredients are listed in the protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with any (serious and non-serious) Adverse Events. | 85 days
  Safety (I)
Number of Participants with abnormal laboratory values. | 85 days
  Safety (II)
Number of Participants with vital sign abnormalities. | 85 days
  Safety (III)
Number of Participants with Adverse Events assessed by 12- lead electrocardiograms (ECGs) | 85 days
  Safety (IV)

CONTACTS AND LOCATIONS:
Overall Officials: Katriina Peltola, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Tuomo Alanko, MD, PhD, Principal Investigator — Docrates Cancer Center
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki, Uusima
  - Docrates Cancer Center, Helsinki, Uusima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clubb JHA, Pakola SA, Joenvaara S, Kudling TV, Tohmola T, Arias V, Jirovec E, van der Heijden M, Quixabeira DCA, Pasanen A, Haybout L, Ojala N, Basnet S, Eleuteri A, Ferrero JD, Hirvenoja S, Svane IM, Maenpaa J, Jalkanen K, Block MS, Alanko T, Monberg T, Zahraoui S, Gronberg-Vaha-Koskela S, Salmelin N, Kistler C, Havunen R, Sorsa S, Manuel Dos Santos J, Cervera-Carrascon V, Kanerva A, Hemminki O, Renkonen R, Hemminki A. Dyslipidemia-associated natural IgM improves oncolytic virus TILT-123 efficacy through antibody-dependent enhancement in solid tumors. Mol Ther. 2026 Jan 20:S1525-0016(26)00020-1. doi: 10.1016/j.ymthe.2026.01.019. Online ahead of print. PMID 41566775
- [Derived] Jirovec E, Quixabeira DCA, Clubb JHA, Pakola SA, Kudling T, Arias V, Haybout L, Jalkanen K, Alanko T, Monberg T, Khammari A, Dreno B, Svane IM, Block MS, Adamo DA, Maenpaa J, Kistler C, Sorsa S, Hemminki O, Kanerva A, Santos JM, Cervera-Carrascon V, Hemminki A. Single intravenous administration of oncolytic adenovirus TILT-123 results in systemic tumor transduction and immune response in patients with advanced solid tumors. J Exp Clin Cancer Res. 2024 Nov 6;43(1):297. doi: 10.1186/s13046-024-03219-0. PMID 39506856